CLINICAL TRIAL: NCT04889976
Title: Psychological Interventions and Transcranial Direct Current Stimulation for the Treatment of Major Depressive Disorder
Brief Title: Portable Transcranial Electrical Stimulation and Internet-Based Behavioral Therapy for Major Depression Study
Acronym: PSYLECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Andre R Brunoni, Associate Professor of the Medical School of the University of Sao Paulo (FMUSP), Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13922419.1.0000.0076; 19/06009-6 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2021-05-10; First posted 2021-05-17 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Major Depressive Disorder; Unipolar Depression
Keywords: major depressive disorder; transcranial electrical stimulation; transcranial direct current stimulation; internet-based behavioral therapy; non-invasive brain stimulation; neuromodulation; home-use transcranial electrical stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: This is a multi-arm, randomized, double-blind, sham-controlled clinical trial with digital features, using portable transcranial electrical stimulation (ptES) and internet-based behavioral therapy (iBT) for major depressive disorder (MDD). The aims of this study are to evaluate the efficacy, safety, tolerability and usability of (1) active ptES + active iBT ("double-active"), (2) active ptES + sham iBT ("ptES-only"), and (3) sham ptES + sham iBT ("double-sham"), in adults with MDD, with a Hamilton Depression Rating Scale - 17 item version (HDRS-17) score ≥ 17 at baseline, during 6 weeks.
Who Masked: Participant, Investigator
Masking Description: The iBT intervention is performed concomitantly to the ptES session, and consists of an app-based interactive protocol (with a chatbot and online videos), synchronized via bluetooth, to the ptES device. For PSYLECT, the chatbot iBT protocol has been translated from English to Portuguese, and all iBT videos are either presented with Portuguese subtitles, or in the case of meditation videos (which allow participants to close their eyes), have been dubbed to Portuguese. Further details about active and sham iBT sessions are not described in this platform to avoid breaking the blinding of future participants enrolled in this study, with means of access to this platform. The complete details will be provided when the study results are published or upon reasonable request.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Double-active (Experimental): Active portable transcranial electrical stimulation (ptES) and active internet-based behavioral therapy (iBT).
  Interventions: Device: Double Active: Active portable transcranial stimulation (ptES) and active internet-based behavioral therapy (iBT)
- ptES-only (Active Comparator): Active portable transcranial electrical stimulation (ptES) and sham internet-based behavioral therapy (iBT).
  Interventions: Device: ptES-only: Active portable transcranial stimulation (ptES) and sham internet-based behavioral therapy (iBT)
- Double-sham (Sham Comparator): Sham portable transcranial electrical stimulation (ptES) and sham internet-based behavioral therapy (iBT).
  Interventions: Device: Double-sham: Sham portable transcranial stimulation (ptES) and sham internet-based behavioral therapy (iBT)

INTERVENTIONS:
Device: Double Active: Active portable transcranial stimulation (ptES) and active internet-based behavioral therapy (iBT) — ptES is delivered by the Flow device (Flow Neuroscience, Malmö, Sweden), consisting of a one-size-fits-all, transcranial direct current stimulation (tDCS) headset with circular electrodes (area = 22.9cm2). The anode is positioned over the left prefrontal cortex, and the cathode over the right prefrontal cortex. Current strength is set at 2mA (current density = 0.087mA/cm2) for 30 minutes, daily for 5 continuous days (with a 2-day pause) for the first 3 weeks, with twice-weekly sessions for the following 3 weeks (total of 21 sessions in 6 weeks). Active iBT consists of a smartphone app with an electronic therapist-avatar. The iBT sessions are delivered concomitantly to the tDCS sessions (the tDCS device connects via bluetooth to the participant's smartphone app).
  Arms: Double-active
Device: ptES-only: Active portable transcranial stimulation (ptES) and sham internet-based behavioral therapy (iBT) — ptES is delivered by the Flow device (Flow Neuroscience, Malmö, Sweden), consisting of a one-size-fits-all, transcranial direct current stimulation (tDCS) headset with circular electrodes (area = 22.9cm2). The anode is positioned over the left prefrontal cortex, and the cathode over the right prefrontal cortex. Current strength is set at 2mA (current density = 0.087mA/cm2) for 30 minutes, daily for 5 continuous days (with a 2-day pause) for the first 3 weeks, with twice-weekly sessions for the following 3 weeks (total of 21 sessions in 6 weeks). The sham iBT sessions are delivered concomitantly to the active ptES sessions (the ptES device connects via bluetooth to the participant's smartphone app).
  Arms: ptES-only
Device: Double-sham: Sham portable transcranial stimulation (ptES) and sham internet-based behavioral therapy (iBT) — Sham ptES for this trial is delivered by the Flow device (Flow Neuroscience, Malmö, Sweden), consisting of a one-size-fits-all transcranial direct current stimulation (tDCS) headset, with circular electrodes (area = 22.9cm2). The anode is positioned over the left prefrontal cortex, and the cathode over the right prefrontal cortex. The sham protocol consists of a fade-in and fade-out phases of 1mA for 45 seconds, followed by a silent period in between for the remaining 28 1/2 minutes. The sham iBT sessions are delivered concomitantly to the sham ptES sessions (the ptES device connects via bluetooth to the participant's smartphone app).
  Arms: Double-sham

SUMMARY:
First-line treatments for major depressive disorder (MDD), antidepressants and psychotherapy, are associated with refractoriness and discontinuation due to side effects, and logistical burdens, respectively. In this scenario, transcranial electrical stimulation (tES) is nowadays considered effective and safe for MDD, albeit with a modest effect size, and also prone to logistical burdens when performed in external facilities. In this regard, clinical investigation involving portable tES (ptES), and the potentiation of ptES with remotely-delivered psychological interventions, have shown positive, but preliminary, results.

Here, the investigators present the design and rationale of a single-center, multi-arm, randomized, double-blind, sham-controlled clinical trial with digital features, using ptES (ptES) and internet-based behavioral therapy (iBT) for MDD (PSYLECT). This study will evaluate the efficacy, safety, tolerability and usability of (1) active ptES + active iBT ("double-active"), (2) active ptES + sham iBT ("ptES-only"), and (3) sham ptES + sham iBT ("double-sham"), in adults with MDD, with a Hamilton Depression Rating Scale - 17 item version (HDRS-17) score ≥ 17 at baseline, during 6 weeks. No antidepressant washouts will be performed during the trial.

Three co-primary hypotheses are presented: changes in HDRS-17 will be greater in (1) "double-active" compared to "ptES-only", (2) "double-active" compared to "double-sham", and (3) "ptES-only" compared to "double-sham".

The investigators aim to enroll 210 patients (70 per arm). The results of this trial should also offer new insights regarding the feasibility and scalability of combined ptES and iBT for MDD, in the area of digital mental health.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a prevalent, debilitating and chronic mental disorder, characterized by frequent recurrences and resistance to first-line treatments: antidepressants and onsite cognitive-behavioral therapy (CBT) are associated with discontinuation due to side-effects, and logistical burdens, respectively.

Non-invasive brain stimulation techniques (NIBS), such as repetitive transcranial magnetic stimulation (rTMS) and transcranial electrical stimulation (tES) (of which the most widely studied format is transcranial direct current stimulation - tDCS), are considered safe and tolerable interventions for MDD. While rTMS is already approved by the FDA for MDD, it involves daily visits to external facilities and is costly.

tES, on the other hand, albeit having failed to prove non-inferiority to a conventional antidepressant (escitalopram 20mg/day) in a previous trial, is less expensive than rTMS, and portable. Therefore, tES could be suitable for home-use under remote supervision by trained clinical staff, especially as an add-on intervention for MDD. In this scenario, recent pilot trials have suggested a possible combined effect of tES with psychological interventions, based on a mechanism known as "functional targeting", that is, using two or more interventions to engage the same brain area of interest.

The PSYLECT study is a parallel, 3-arm, randomized, double-blind, sham-controlled, single-center clinical trial, with digital features, devised to assess the efficacy, tolerability, safety and usability of: (1) active portable tES (ptES) + active internet-based behavioral therapy (iBT) ("double active"), (2) active ptES + sham iBT ("ptES-only"), and (3) sham ptES + sham iBT ("double-sham"), for the treatment of MDD, in adults, during 6 weeks.

The investigators will enroll 210 adult patients (70 per arm) diagnosed with MDD per DSM-5 criteria, regardless of being in treatment with conventional antidepressants, to receive either: "double-active", "ptES-only" or "double-sham", during 6 weeks.

The use of sham (placebo) is necessary in order to better estimate the combined active treatment effect, but patients will be invited to receive the active treatments at endpoint, in an open-label 6-week, crossover phase, if they were previously randomized to receive "double-sham", and did not display response at endpoint (defined ≥ 50% reduction in depressive symptoms). Furthermore, patients who were randomized to "double-active" or "ptES-only" and display response at endpoint, will be invited to participate in a maximum 6-month open-label follow-up phase (including those patients that respond at the end of the cross-over period). However, participants who were randomized to "ptES-only", but do not achieve response, will not be eligible for open-label follow-up, as it is unlikely they would profit from a continuation.

The study has received approval by the Ethics Committee of the University of Sao Paulo, in accordance with the Declaration of Helsinki guidelines. Prior to enrollment, participants and researchers will receive and jointly sign an informed consent document.

In this study, 3 co-primary hypotheses are presented: (1) changes in depression scores in the Hamilton Depression Rating Scale 17-item version (HDRS-17), from baseline to endpoint, will be larger in the "double active" compared to the "ptES-only" arm; (2) changes in depression scores (HDRS-17), from baseline to endpoint, will be larger in the "double active" compared to the "double-sham" arm; and (3) changes in depression scores (HDRS-17), from baseline to endpoint, will be larger in the "ptES-only" as compared to the "double-sham" arm.

The secondary hypotheses are that: (1) changes in depression scores will be larger in "double-active" compared to "ptES-only", in "double-active" compared to "double-sham", and "ptES-only" compared to "double-sham" arms, using additional depression-rating scales; (2) response (defined as ≥ 50% reduction in HDRS-17) and remission (defined as HDRS-17 ≤ 7) will be larger in "double active" versus "ptES-only", "double-active" versus "double-sham", and "ptES-only" versus "double sham" arms; (3) reduction in anxiety symptom scores will be greater in "double-active" compared "ptES-only", "double-active" compared to "double-sham", and "ptES-only" compared to "double-sham"; (4) the clinical usability of the "double active" protocol will be regarded as (very) easy by ≥ 80% of recipients, according to a Likert scale; (5) all three protocols will be equally safe and tolerable, according to the tDCS Adverse Events Survey.

Prior to performing online home-based sessions, participants will receive proper onsite training with the ptES device and iBT app, and from then on, will have remote access to the investigators through a phone line and email for questions and management of adverse events. In this case, patients can be redirected to the research institution's clinical facilities (including its emergency departments), in case of clinical and/or psychiatric adverse events which are deemed to need onsite evaluation and follow-up. The aforementioned clinical facilities are situated at the Clinics and University Hospitals of the University of Sao Paulo, Brazil, which are, respectively, tertiary and secondary care centers, and reference public hospitals in the Sao Paulo city area.

The ptES devices used in this trial are manufactured by Flow Neuroscience (Malmö, Sweden), and consist of a one-size-fits-all headset with circular electrodes, with the anode positioned over the left prefrontal cortex and the cathode over the right prefrontal cortex. The device comes with a set of 21 sealed, saline-humidified disposable sponges, an electrical charger, and has pre-set and fixed stimulation parameters. This device has been previously tested by the investigators in a computer-modeling procedure, with simulations displaying adequate electrical field strength and distribution in prefrontal brain areas of interest (ie, dorsolateral prefrontal cortex). Furthermore, the Flow device has been approved in the United Kingdom, European Union and Brazil (National Agency of Sanitary Vigilance, ANVISA), for home-use in patients with MDD.

The investigators' team will consist of 2 separate groups: (1) unblinded "session supervisors", who will offer an initial onsite training session to participants and will be available remotely for supervised guidance for the following online home-based sessions; (2) blinded clinical evaluators, who will evaluate participants online weekly until study endpoint, while being able to refer patients to onsite evaluation, as deemed necessary.

For data collection, the investigators will use REDCap (Research Electronic Data Capture), created at Vanderbilt University (Tennessee, USA) with NIH support. REDCap is a free-source software, that works in offline and online modes and runs on tablets, smartphones and computers, and was designed to build and manage online surveys and databases, replacing paper notebooks. It also has tools that allow dynamic data management and data quality examination. REDCap can be installed in a variety of environments for compliance with such standards as HIPAA, 21 CFR Part 11, FISMA (low, moderate, high), Brazlian regulations (LGPD) and international standards.

Periodically, the data will be exported and saved offline in password-protected external HDs and flash drives. REDCap access will be restricted using individual usernames and passwords. No user will have permission to modify or export the data (except for generating security copies) during the trial. If data edition is necessary (e.g., incorrect input), a new data version will be generated. All changes in the data will be reported.

For data management and quality control, the investigators hired an information technology (IT) specialist for technical support in the project. Data will be coded according to a previously developed data dictionary. Quality of data collection will be monitored by random data quality checks for consistency (e.g., depression scores compatible in different scales) and completeness (absence or few cases of missing data). The investigators will also have access to an online dashboard, that remotely monitors participant adherence to study protocol.

If unblinding is necessary, the PI holds special codes for the procedure, while having to specify the reason for unblinding, which are: an increase ≥ 25% from baseline scores on the Hamilton Depression Rating Scale-HDRS (17-item version) on 2 consecutive clinical evaluations, development of suicidal ideation, serious clinical and psychiatric adverse events, development of hypo(mania) and/or psychotic symptoms, low adherence (missing 2 clinical evaluations or failing to comply with at least 75% of tDCS sessions at home) or patient consent withdrawal.

For the sample size calculations, baseline depression scores and standard deviation (SD) of 25 (±5) on the HDRS-17 were used, distributed equally between groups, based on previous studies. Furthermore, the investigators consider that: (1) placebo effects in the double-sham arm will impact baseline depression scores equal to 1 effect size (ES) in SD units (ES = difference in mean change divided by SD); (2) the "ptES-only" arm will have the same placebo effects present in the double-sham arm (ES = 1), plus a treatment response of ES = 0.4; and, (3) the "double-active" arm will have placebo effects (ES = 1) plus a larger response of ES = 0.8. Therefore, probable endpoint scores of 20, 18 and 16 were used, for "double-sham", "ptES-only" and "double-active", respectively. The effect sizes were also chosen based on the results from previous trials, and considering that tDCS and online behavioral therapies have small to moderate effect sizes.

Sample size per arm was calculated based on the smallest detectable group difference (ES tDCS vs. combination = -0.4, ES sham vs. tDCS = -0.4). Significance levels were Bonferroni corrected for 3-way pairwise comparisons (α = 0.05/3) to control family-wise error rate, while still allowing for more anti-conservative adjustment in the final analysis. Dropouts were assumed to be monotonically increasing (Weibull) and equally distributed between treatment arms. The investigators obtained a total n = 210 participants, assuming a 10% attrition rate (therefore, 70 persons per arm).

Results will be considered statistically significant if a two-sided p<0.0167 (Bonferroni-corrected) is obtained. For the analysis of the co-primary outcomes, a linear mixed-effect model (LLM) will be employed, using a first order regressive covariance structure, which includes all observed variables without the need of imputing missing data. The dependent variable is score change on the HDRS-17. Independent variables are time (all observations until week 6), and group ("double-active", "ptES-only" and "double-sham"). The investigators will test the statistical significance between the pairwise comparisons per our primary hypotheses. The investigators will employ an intention-to-treat (ITT) approach. For the analysis of the secondary outcomes, linear mixed-effects models will be employed analogically to the analysis for the primary outcomes. Binary outcomes (response and remission) will be modeled using mixed logistic regression at each time-point. Improvement in other depressive domains will be evaluated using the same linear hierarchical models described.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder (MDD) per DSM-5 criteria
* Hamilton Rating Scale (17-item version)-HDRS score ≥ 17 at baseline
* Years of education ≥ 8
* Having access to a smartphone with internet access at home
* Treatment refractoriness ≤ 3 antidepressants, at optimal doses and for appropriate duration
* No contraindications for tDCS (i.e., metallic plates on the head, brain devices, cochlear implants, cardiac pacemakers)
* No suicidal ideation with planning, or attempted suicide, in the 4 weeks prior to baseline

Exclusion Criteria:

* Other psychiatric diagnoses (i.e., schizophrenia, schizoaffective disorder, bipolar disorder, obsessive compulsive disorder, attention-deficit and hyperactivity disorder, personality disorders, substance dependence and/or abuse disorders). Obs.: Anxiety disorders, as a comorbidity, will not be an exclusion criterium.
* Suspected or confirmed pregnancy
* Lactation
* Severe clinical or neurological conditions, including Post-Acute Sequelae of COVID-19
* Depressive symptoms better explained by other clinical conditions (i.e., hypothyroidism, anemia) or other psychiatric disorders.
* Use of benzodiazepines > 10mg diazepam or diazepam-equivalent per day

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale scores (17-item version) between "double active" and "ptES-only" | Week 0 (baseline) and Week 6.
  Clinician-administered depression assessment scale. Score range = 0 - 52 (higher scores mean worse outcome).
Change in Hamilton Depression Rating Scale scores (17-item version) between "double active" and "double-sham" | Week 0 (baseline) and Week 6.
  Clinician-administered depression assessment scale. Score range = 0 - 52 (higher scores mean worse outcome).
Change in Hamilton Depression Rating Scale scores (17-item version) between "ptES-only" and "double-sham" | Week 0 (baseline) and Week 6.
  Clinician-administered depression assessment scale. Score range = 0 - 52 (higher scores mean worse outcome).

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale scores (17-item version) | Weeks 0, 2, 3, 4 and 6.
  Clinician-administered depression assessment scale. Score range = 0 - 52 (higher scores mean worse outcome).
Change in Montgomery-Asberg Depression Rating Scale scores (MADRS) | Weeks 0, 2, 3, 4 and 6.
  Clinician-administered depression assessment scale. Score range = 0 - 60 (higher scores mean worse outcome).
Change in Beck Depression Inventory - II scores (BDI - II) | Weeks 0, 2, 3, 4 and 6.
  Self-report depressive symptoms inventory. Score range = 0 - 63 (higher scores mean worse outcome).
Change in Hamilton Anxiety Rating Scale scores (HAM-A) | Weeks 0, 3 and 6.
  Clinician-administered anxiety assessment scale. Score range = 0 - 30 (higher scores mean worse outcome).
Change in Clinical Global Impression Rating Scale (Severity of Illness) scores (CGI-S) | Weeks 0 and 6.
  Clinician-administered scale that measures illness-severity. Score range = 0 - 7 (higher scores mean worse outcome).
Clinical Global Impression Rating Scale (Global Improvement) score (CGI-I) | Week 6.
  Clinician-administered scale that measures global improvement to treatment. Score range = 0 - 7 (higher scores mean worse outcome).
Change in Young Mania Rating Scale (YMRS) scores | Weeks 2, 3, 4 and 6.
  Clinician-administered scale that measures hypomania/mania symptoms. Score range = 0 - 60 (higher scores mean worse outcome).
Change in Positive and Negative Affect Schedule scores (PANAS) | Weeks 0, 3 and 6.
  Self-report questionnaire to measure both positive and negative affect. Positive Affect Score: scores can range from 10 - 50, with higher scores representing higher levels of positive affect (better outcome). Negative Affect Score: scores can range from 10 - 50, with higher scores representing higher levels of negative affect (worse outcome).
Change in State-Trait Anxiety Inventory scores (STAI-T and STAI-S) | Weeks 0, 3 and 6.
  Self-report measures of state and trait anxiety. The range of possible scores for each subscale (STAI-T and STAI-S) varies from a minimum score of 20 to a maximum score of 80, with higher scores meaning worse outcome.
Change in Device usability Likert scale scores | Weeks 1, 2, 3, 4, 5 and 6.
  Self-report visual analog device usability scale. Score range = 0 - 100. Higher scores mean better outcome.
Change in tDCS Adverse Event Questionnaire scores | Weeks 1, 2, 3, 4, 5 and 6.
  Self-report tDCS adverse event questionnaire, with quantitative symptom intensity and association scores. Scores for the symptom intensity subscale range from 16 - 64, with higher scores meaning worse outcome; scores on the symptom association subscale range from 16 - 80, with higher scores meaning worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Institute of Psychiatry, HC-FMUSP, São Paulo, São Paulo
  - Hospital Universitário - USP, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sathappan AV, Luber BM, Lisanby SH. The Dynamic Duo: Combining noninvasive brain stimulation with cognitive interventions. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Mar 8;89:347-360. doi: 10.1016/j.pnpbp.2018.10.006. Epub 2018 Oct 9. PMID 30312634
- [Background] Brunoni AR, Moffa AH, Sampaio-Junior B, Borrione L, Moreno ML, Fernandes RA, Veronezi BP, Nogueira BS, Aparicio LVM, Razza LB, Chamorro R, Tort LC, Fraguas R, Lotufo PA, Gattaz WF, Fregni F, Bensenor IM; ELECT-TDCS Investigators. Trial of Electrical Direct-Current Therapy versus Escitalopram for Depression. N Engl J Med. 2017 Jun 29;376(26):2523-2533. doi: 10.1056/NEJMoa1612999. PMID 28657871
- [Background] Brunoni AR, Valiengo L, Baccaro A, Zanao TA, de Oliveira JF, Goulart A, Boggio PS, Lotufo PA, Bensenor IM, Fregni F. The sertraline vs. electrical current therapy for treating depression clinical study: results from a factorial, randomized, controlled trial. JAMA Psychiatry. 2013 Apr;70(4):383-91. doi: 10.1001/2013.jamapsychiatry.32. PMID 23389323
- [Background] Segrave RA, Arnold S, Hoy K, Fitzgerald PB. Concurrent cognitive control training augments the antidepressant efficacy of tDCS: a pilot study. Brain Stimul. 2014 Mar-Apr;7(2):325-31. doi: 10.1016/j.brs.2013.12.008. Epub 2013 Dec 19. PMID 24486425
- [Background] Brunoni AR, Boggio PS, De Raedt R, Bensenor IM, Lotufo PA, Namur V, Valiengo LC, Vanderhasselt MA. Cognitive control therapy and transcranial direct current stimulation for depression: a randomized, double-blinded, controlled trial. J Affect Disord. 2014 Jun;162:43-9. doi: 10.1016/j.jad.2014.03.026. Epub 2014 Mar 27. PMID 24767004
- [Background] Razza LB, Afonso Dos Santos L, Borrione L, Bellini H, Branco LC, Cretaz E, Duarte D, Ferrao Y, Galhardoni R, Quevedo J, Simis M, Fregni F, Correll CU, Padberg F, Trevizol A, Daskalakis ZJ, Carvalho AF, Solmi M, Brunoni AR. Appraising the effectiveness of electrical and magnetic brain stimulation techniques in acute major depressive episodes: an umbrella review of meta-analyses of randomized controlled trials. Braz J Psychiatry. 2021 Sep-Oct;43(5):514-524. doi: 10.1590/1516-4446-2020-1169. PMID 33111776
- [Background] Borrione L, Suen PJC, Razza LB, Santos LAD, Sudbrack-Oliveira P, Brunoni AR. The Flow brain stimulation headset for the treatment of depression: overview of its safety, efficacy and portable design. Expert Rev Med Devices. 2020 Sep;17(9):867-878. doi: 10.1080/17434440.2020.1813565. Epub 2020 Sep 7. PMID 32820677
- [Background] Charvet LE, Shaw MT, Bikson M, Woods AJ, Knotkova H. Supervised transcranial direct current stimulation (tDCS) at home: A guide for clinical research and practice. Brain Stimul. 2020 May-Jun;13(3):686-693. doi: 10.1016/j.brs.2020.02.011. Epub 2020 Feb 10. PMID 32289698
- [Background] Alonzo A, Fong J, Ball N, Martin D, Chand N, Loo C. Pilot trial of home-administered transcranial direct current stimulation for the treatment of depression. J Affect Disord. 2019 Jun 1;252:475-483. doi: 10.1016/j.jad.2019.04.041. Epub 2019 Apr 10. PMID 31005790
- [Background] Brunoni AR, Sampaio-Junior B, Moffa AH, Aparicio LV, Gordon P, Klein I, Rios RM, Razza LB, Loo C, Padberg F, Valiengo L. Noninvasive brain stimulation in psychiatric disorders: a primer. Braz J Psychiatry. 2019 Jan-Feb;41(1):70-81. doi: 10.1590/1516-4446-2017-0018. Epub 2018 Oct 11. PMID 30328957
- [Derived] Borrione L, Cavendish BA, Aparicio LVM, Luethi MS, Goerigk S, Ramos MRF, Moran NKS, Carneiro AM, Valiengo L, Moura DO, de Souza JP, Batista MP, Aparecida da Silva V, Klein I, Suen P, Gallucci-Neto J, Padberg F, Razza LB, Vanderhasselt MA, Lotufo PA, Bensenor IM, Fregni F, Brunoni AR. Home-Use Transcranial Direct Current Stimulation for the Treatment of a Major Depressive Episode: A Randomized Clinical Trial. JAMA Psychiatry. 2024 Apr 1;81(4):329-337. doi: 10.1001/jamapsychiatry.2023.4948. PMID 38170541
- [Derived] Borrione L, Cirillo PC, Aparicio LV, Cavendish BA, Valiengo L, Moura DO, de Souza JP, Luethi MS, Klein I, Bariani B, Gallucci-Neto J, Suen P, Padberg F, Goerigk S, Vanderhasselt MA, De Deng Z, O'Shea J, Lotufo PA, Bensenor IM, Brunoni AR. A study protocol for an ongoing multi-arm, randomized, double-blind, sham-controlled clinical trial with digital features, using portable transcranial electrical stimulation and internet-based behavioral therapy for major depression disorders: The PSYLECT study. Expert Rev Neurother. 2022 Jun;22(6):513-523. doi: 10.1080/14737175.2022.2083959. Epub 2022 Jun 8. PMID 35642516
- See also: Information site of the Interdisciplinary Service of Neuromodulation Department of the Institute of Psychiatry of the University of Sao Paulo Medical School (research and assistance) — http://www.sin.org.br